CLINICAL TRIAL: NCT01701713
Title: Safety Study of Transcranial Direct Current Stimulation in Aphasia Therapy in Acute and Post-acute Stroke
Brief Title: TDCS in Acute Stroke
Acronym: TDCS-aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Brandenburg Klinik, Bernau, Germany (Unknown); University of Potsdam (Other)
Responsible Party: Principal Investigator, Gerhard Jan Jungehuelsing, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TDCS_CSB-Brandenburg; EA4/109/08 (Other: Charité Ethics Committee)
Record Dates: First submitted 2012-09-26; First posted 2012-10-05 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Stroke
Keywords: TDCS; STROKE; APHASIA; NAMING
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDCS - DKI ED2011 (Experimental): TDCS with DKI ED2011 session is followed by a behavioral naming therapy with different cues
  Interventions: Device: DKI ED2011
- Sham-TDCS (Sham Comparator): Sham-TDCS session is followed by a behavioral naming therapy with different cues
  Interventions: Device: Sham-TDCS

INTERVENTIONS:
Device: DKI ED2011
  Arms: TDCS - DKI ED2011
Device: Sham-TDCS
  Arms: Sham-TDCS

SUMMARY:
The purpose of this study is to determine the safety of transcranial direct current stimulation in aphasia therapy in acute and post-acute stroke.

DETAILED DESCRIPTION:
TDCS has been shown to have a positive effect on clinical outcome in both motor rehabilitation and aphasia treatment in chronic aphasic patients. In healthy subjects the method sped up reaction times in naming and language learning tasks. In TDCS a weak current is applied to the subjects head increasing excitatory activity which might lead to improved brain function.

ELIGIBILITY:
Inclusion Criteria:

* first media stroke
* language impairment
* informed consent
* right handedness
* NIHSS < 20

Exclusion Criteria:

* previous Epilepsy oder epileptogenic events
* epilepsy typical elements in EEG
* hypersensitive skin (head)
* metal implants (head)
* pace maker or other electronic implants
* previous head/brain surgery
* medication reducing seizure threshold
* previous psychiatric events

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
skin irritation | 2 months

SECONDARY OUTCOMES:
Improved language | 2 months
  improved picture naming

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard J Jungehuelsing, MD, Principal Investigator — Center for Stroke Research Berlin (CSB), Charité; Michael Joebges, Prof. MD, Principal Investigator — Brandenburgklinik Bernau
Locations (2):
- Germany (2):
  - Brandenburg Klinik Bernau, Bernau bei Berlin, Brandenburg
  - Charité, Campus Benjamin Franklin, Dep. of Neurology, Berlin, State of Berlin